CLINICAL TRIAL: NCT02041858
Title: Effect of Altered Alarm Settings on Patient Adverse Events and Alarm Signal Frequency: A Randomized Controlled Trial Feasibility Study
Brief Title: Effect of Altered Alarm Settings on Patient Adverse Events and Alarm Signal Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Julius Cuong Pham, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00079765
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Physiologic Monitoring; Alarms
Keywords: Alarms; Physiologic Monitoring; Critical Care; Alarm fatigue; Adverse Events
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control arm with organizational-based alarm parameter settings
- Altered Alarm Settings (Experimental): Altered set of alarm parameter settings.
  Interventions: Other: Altered Alarm Settings

INTERVENTIONS:
Other: Altered Alarm Settings — An altered set of alarm parameter settings
  Arms: Altered Alarm Settings

SUMMARY:
Alarm fatigue, a lack of response to an alarm due to desensitization, is a national problem. The problem of alarm desensitization is multifaceted and is related to a high false alarm rate, poor positive predictive value, lack of alarm standardization and the large number of medical devices with built in alarms in use today. Cardiac monitor alarms are intended to notify the healthcare practitioner that a clinical crisis is imminent. However, hundreds of physiologic monitor alarms occur on monitored units each day. As a result, practitioners are highly vulnerable to alarm fatigue which has resulted in serious harm to patients and death due to staff inattention from alarm signal desensitization. Research indicates that 80-99.4% of monitor alarms are false or clinically insignificant. Alarm hazards is the number one medical device technology hazard of 2012 and has been listed by ECRI (Emergency Care Research Institute) among the top 3 medical device hazards for the past three years (ECRI, 2011). Delivering actionable alarm information to care providers is challenging given the significant number of false alarms.

Ideally, alarms should activate for events in greatest need of clinical attention without increasing the risk of adverse patient outcomes. This is not the case with current monitoring technology which is designed for high sensitivity and low specificity. Practitioners must use clinical intuition for determining how conservatively alarms should be set to be most useful. There is no research evidence to support how best to set alarms without affecting patient outcomes.

Quality improvement studies performed at The Johns Hopkins Hospital have demonstrated that the frequency of alarm signals can be reduced by more than 50% through an altered set of alarm parameters. This reduction in alarm signals has lead to an increase awareness of alarms that do occur as well as create a quieter, healing environment for patients. Although this change was not associated with a "noticeable" increase in adverse patient events, this important outcome was not rigorously studied.

The specific aims of this pilot study is to determine if decreasing the number of alarms by using an altered set of alarm parameters has an effect on patient outcomes in an intensive care unit.

This project may have a significant impact on patient safety. A decrease in noise at the bedside may result in less distraction to caregivers and may have a positive effect on patient recovery. It is expected that the altered set of monitor default parameters will result in a decrease in audible alarms without increasing clinically significant adverse patient events.

ELIGIBILITY:
Inclusion Criteria: All patients who are in the Coronary Care Unit and able to provide consent during the collection time period will be considered for inclusion. This unit consists of adult patients with a primary cardiac etiology for their illness. The vast majority of these patients are either there for coronary artery disease or congestive heart failure.

Exclusion Criteria: Patients who are unable to provide consent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinically significant adverse events | 1 day
  A variety of clinically significant events were assessed while subjects were on the protocol

SECONDARY OUTCOMES:
Alarm Signals | 1 day
  The number of alarm signals were assessed while the subject was on the protocol.
Alarm-triggered interventions | 1 day
  The number and type of alarm-triggered interventions were assessed while the patient was on the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Julius C Pham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cvach M. Monitor alarm fatigue: an integrative review. Biomed Instrum Technol. 2012 Jul-Aug;46(4):268-77. doi: 10.2345/0899-8205-46.4.268. PMID 22839984
- [Background] Lawless ST. Crying wolf: false alarms in a pediatric intensive care unit. Crit Care Med. 1994 Jun;22(6):981-5. PMID 8205831
- [Background] Tsien CL, Fackler JC. Poor prognosis for existing monitors in the intensive care unit. Crit Care Med. 1997 Apr;25(4):614-9. doi: 10.1097/00003246-199704000-00010. PMID 9142025
- [Background] Chambrin MC, Ravaux P, Calvelo-Aros D, Jaborska A, Chopin C, Boniface B. Multicentric study of monitoring alarms in the adult intensive care unit (ICU): a descriptive analysis. Intensive Care Med. 1999 Dec;25(12):1360-6. doi: 10.1007/s001340051082. PMID 10660842
- [Background] Atzema C, Schull MJ, Borgundvaag B, Slaughter GR, Lee CK. ALARMED: adverse events in low-risk patients with chest pain receiving continuous electrocardiographic monitoring in the emergency department. A pilot study. Am J Emerg Med. 2006 Jan;24(1):62-7. doi: 10.1016/j.ajem.2005.05.015. PMID 16338512
- [Background] Siebig S, Kuhls S, Imhoff M, Langgartner J, Reng M, Scholmerich J, Gather U, Wrede CE. Collection of annotated data in a clinical validation study for alarm algorithms in intensive care--a methodologic framework. J Crit Care. 2010 Mar;25(1):128-35. doi: 10.1016/j.jcrc.2008.09.001. Epub 2009 Jan 17. PMID 19327311